CLINICAL TRIAL: NCT06267937
Title: Hip Fractures in Chile: Implications for Public Health Policy and Healthcare Delivery
Status: Completed | Type: Observational
Sponsor: University of Chile (Other)
Collaborators: Instituto Sistemas Complejos de Ingeniería, Universidad de Chile, Santiago, Chile (Unknown)
Responsible Party: Principal Investigator, maximiliano barahona vasquez, Associate proffesor, University of Chile
Other Study IDs: 101
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hip fracture: patients that were diagnosed with a hip fracture between 2012 and 2017
  Interventions: Procedure: Access to surgery; Other: type of intitution

INTERVENTIONS:
Procedure: Access to surgery — access to surgery after hip fracture
Other: type of intitution — public or private health care facility

SUMMARY:
Hip fractures in individuals aged 60 and above pose significant challenges in terms of morbidity, mortality, and healthcare costs. While countries like the United Kingdom and Australia have optimized their healthcare systems for timely management of hip fractures, the situation in Chile presents distinct challenges due to its mixed healthcare system. This study aims to assess survival rates following hip fractures in Chile and identify associated risk factors using national databases from 2012 to 2018. A comprehensive analysis of 35,520 patients revealed that factors such as age, type of health insurance, access to surgery, and treatment in public hospitals significantly influence mortality rates after hip fractures. The study found that patients with hip fractures experience lower 5-year survival rates compared to the general population, particularly when affiliated with public insurance and treated in public institutions. Modifiable factors like delayed surgery and prolonged hospital stays contribute to increased mortality rates. The findings underscore the urgent need for optimized public health policies and healthcare delivery systems to enhance outcomes for hip fracture patients in Chile.Hip fractures in individuals aged 60 and above pose significant challenges in terms of morbidity, mortality, and healthcare costs. While countries like the United Kingdom and Australia have optimized their healthcare systems for timely management of hip fractures, the situation in Chile presents distinct challenges due to its mixed healthcare system. This study aims to assess survival rates following hip fractures in Chile and identify associated risk factors using national databases from 2012 to 2018.

ELIGIBILITY:
Inclusion Criteria:

All patients in the national database between 2012 and 2017 which his principal was hip fracture. Diagnoses are classified using the International Classification of Diseases, 10th Revision (ICD-10) codes. A search was conducted for codes S72.0 (head and neck fracture of the femur), S72.1 (pertrochanteric fracture), and S72.2 (subtrochanteric fracture of the femur).

Exclusion Criteria:

missing IDs ID with inconsistent socio-demographic information. Patients with primary diagnosis of hip fracture that underwent surgery but the national code surgery was not one of the following: : 2104128, 2104129, 2104131, 2104132, 2104135, 2104228, 2104229 and 2104231

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The chilean national database of hospital discharge and the chilean death registry from 2012 to 2018 were used. , The date of death was recorded for the 35,520 patients who had deceased; otherwise, they are classified as alive as of the current date. We remark that the national discharge and death databases use the same patient IDs, and therefore, we can easily identify those patients who have died during the period under analysis. We notice that we have used the hospital discharge database up to 2017 to have at least one year of follow-up for patients after a hip fracture.
Sampling Method: Non-Probability Sample
Enrollment: 46380 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
survival after hip fracture | one to five years after the hip fracture
  survival after hip fracture

CONTACTS AND LOCATIONS:
Overall Officials: Susana Mondschein, PhD, Study Chair — University of Chile
Locations (1):
- hospital Clinico Universidad de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Yes
Both National regestries are free access, nevertheless, the raw data will be made available after publication.
Supporting Information: Study Protocol
Time Frame: after publication, until 10 years.